CLINICAL TRIAL: NCT03071172
Title: Clinical Study of Recombinant Human Follitropin for Injection Assisted in Controlled Ovarian Hyperstimulation Assisted IVF-ET
Brief Title: Clinical Study of Recombinant Human Follitropin for Injection Assisted in COH Assisted IVF-ET
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Peking University Third Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Women's Hospital School Of Medicine Zhejiang University (Other); Xiangya Hospital of Central South University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GenSci 067 CT
Record Dates: First submitted 2017-02-20; First posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-02

CONDITIONS: Ovarian Hyperstimulation Syndrome
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Triptorelin Pamoate; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Human Follitropin (Experimental): Experimental group (domestic rhFSH, powder for injection, 5.5μg (75IU)/vial, initial dose 150-225IU/d, subcutaneous injection, adjust the dose according to ovarian reactivity after 5-7 days of injections, once a day until the HCG trigger day.
  Interventions: Drug: Triptorelin for Injection; Drug: Recombinant Human Choriogonadotropin alfa Solution for Injection; Drug: Progesterone Soft Capsules
- Gonal-F (Active Comparator): Positive control group (imported rhFSH, powder for injection, 5.5μg (75IU)/vial, initial dose 150-225IU/d, subcutaneous injection, adjust the dose according to ovarian reactivity after 5-7 days of injections, once a day until the HCG trigger day.
  Interventions: Drug: Triptorelin for Injection; Drug: Recombinant Human Choriogonadotropin alfa Solution for Injection; Drug: Progesterone Soft Capsules

INTERVENTIONS:
Drug: Triptorelin for Injection — Drugs for IVF-ET (in vitro fertilization and embryo transfer).
  Other Names: Gonadotropin releasing hormone agonists
Drug: Recombinant Human Choriogonadotropin alfa Solution for Injection — Drugs for IVF-ET (in vitro fertilization and embryo transfer).
Drug: Progesterone Soft Capsules — Drugs for IVF-ET (in vitro fertilization and embryo transfer).

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of domestic recombinant human follicle stimulating hormone (rhFSH) stimulating ovarian to promote follicular development before assisted reproductive technology, which was non-inferiority than that of the imported rhFSH.

ELIGIBILITY:
Inclusion Criteria:

* Age is more than 20 years old and less than 39 years old, married.
* Applicable for ART controlled ovarian hyperstimulation, such as IVF/ET, ICSI, GIFT, ZIFT and so on.
* Regular menstrual cycle (25-35 days).
* 18kg/m2≤BMI<30kg/m2.
* The level of basic serum FSH <10IU / L in the 2nd-5th days of the menstrual cycle, the luteinizing hormone, estradiol and progesterone levels were normal.
* The screening period or recent three months of vaginal ultrasound examination showed that the shape of bilateral ovarian and uterine size were normal and 5 ≤ number of basal antral follicle in unilateral ovarian <10, and follicular diameter <10 mm.
* The in vitro fertilization and embryo transfer (IVF/ET) and (or) intracytoplasmic sperm injection (ICSI) technology were less than three times used prior to the reproductive treatment (provide copies of previous cases).
* Volunteer to participate and sign informed consent.

Exclusion Criteria:

* There are high risk of ovarian hyperstimulation syndrome (OHSS), such as the subject who has high response to gonadotropin in the previous ovarian hyperstimulation cycle, polycystic ovary syndrome (PCOS), the subject who has severe OHSS cancellation cycle.
* Affect the outcome of pregnancy-related diseases (any one): untreated hydrosalpinx, untreated uterine polyps, untreated uterine infection, stage Ⅲ ~ IV endometriosis, ovarian cyst> 4cm , uterine fibroids diameter> 4cm, pelvic benign tumor> 4cm, pituitary tumors and malignant tumors of tissues and organs.
* The subject has abnormal uterine bleeding.
* Affect pregnancy-related endocrine and metabolic diseases (any one): hyperprolactinemia, thyroid disease (including hyperthyroidism, hypothyroidism), hyperandrogenism, adrenal dysfunction (including adrenal hyperfunction, adrenal cortical dysfunction).
* The subject has severe liver and kidney dysfunction, which the levels of serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are 2.5 times higher than the upper limit of normal value, and serum creatinine (Cr) and urea nitrogen (BUN) are 2 times higher than the upper limit of normal value.
* Severe heart disease, unstable angina pectoris, heart failure grade Ⅲ above, acute myocardial infarction and/or old myocardial infarction, hypertension diagnosed according to the 2010 edition of the Chinese Hypertension Prevention Guidelines.
* The subject who have contraindications or allergic history for gonadotropin-releasing hormone agonists (GnRH-a), rFSH/human menopausal gonadotropin (hMG), human chorionic gonadotropin (hCG), progesterone drugs.
* Positive HIV or syphilis.
* The subject has alcoholism, smoking, drug abuse, bad drug abuse habits.
* At least one of the spouses has received sperm donor or egg donor or PGD (genetic diagnosis before embryo transfer) and PGS (Preimplantation of embryos before genetic screening)。
* The subject received clomiphene or gonadotropin therapy within 1 month before screening。
* The subject was participated in last three months or are participating in other clinical research。
* Patients with positive serum pregnancy test.
* The investigators considered the subject inappropriate to be enrolled in this study.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
The total number of oocytes obtained during the start-up period | On the days of ovum picking up (hCG trigger 36-38h)
  Routine ova harvest to determine the number of obtained oocytes

SECONDARY OUTCOMES:
The number of follicle-1 | on the day of hCG day
  The number of follicle with diameter more than 18mm
The number of follicle-2 | on the fifth day of rhFSH ovarian stimulation
  The number of follicle with diameter more than 18mm
Number of 2PN oocytes | Collected on the day of embryo transfer day after three days of ovum picking up.
Number of metaphase II oocytes | Collected on the day of embryo transfer day after three days of ovum picking up, which only collected during ICSI cycle.
Number of transferred embryos | Collected on the day of embryo transfer day after three days of ovum picking up.
Number of high quality embryos | Collected on the day of embryo transfer day after three days of ovum picking up.
Fresh cycle embryo implantation | Collected on the day of embryo transfer day after three days of ovum picking up.
rhFSH administered days and vials; administered total dose of rhFSH (IU) | Collected on the day of hCG day.
Serum E2 level | Collected on the day of hCG day.
High quality embryos rate | Collected on the day of embryo transfer day after three days of ovum picking up.
Fertilization rate | Collected on the day of embryo transfer day after three days of ovum picking up.
Fresh cycle embryo implantation rate | Collected between 28-35 days after embryo transfer.
Biochemical pregnancy rate | Collected between 14-16 days after embryo transfer.
Clinical pregnancy rate | Collected between 28-35 days after embryo transfer.
Continuous pregnancy rate | Collected after 12 weeks of embryo transfer.
The number of follicle-3 | on the day of hCG day
  The number of follicle with diameter between 14mm and 18mm.
The number of follicle-4 | on the day of hCG day
  The number of follicle with diameter less than 14mm
Endometrium thickness (mm) | on the day of hCG

CONTACTS AND LOCATIONS:
Overall Officials: Rong Li, Doctor, Principal Investigator — Peking University Third Hospital
Locations (7):
- China (7):
  - The first Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Peking University Third Hospital, Beijing
  - Jiangsu Province Hospital, Nanjing